CLINICAL TRIAL: NCT04805060
Title: A Phase I, Open-label, Dose Escalation Study to Evaluate the Tolerance and Pharmacokinetics of TQB2858 Injection in Subjects With Terminal Malignant Tumor
Brief Title: A Study to Evaluate the Tolerance and Pharmacokinetics of TQB2858 Injection in Subjects With Terminal Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TQB2858-I-01
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Terminal Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2858 injection (Experimental): TQB2858 administered intravenously (IV) once every 3 week
  Interventions: Drug: TQB2858 injection

INTERVENTIONS:
Drug: TQB2858 injection — TQB2858 administered intravenously (IV) on Day 1 of each 21-day. The established dose of TQB2858 is diluted with normal saline [0.9% (w/v) sodium chloride solution], and the infusion time is 60 ± 10 min.

SUMMARY:
This study is a phase I study to evaluate the safety and tolerability of TQB2858 injection in patients with advanced malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced malignancies diagnosed histologically and/or cytologically, where standard treatment has failed or there is no effective treatment;
* Age: 18-75 years old;
* ECOG score: 0 ~ 1;
* Expected survival of more than 3 months;
* The main organs are functioning normally;
* Women of childbearing age must be negative for serum or urine HCG within 7 days prior to study enrollment and must be non-lactating;Patients should agree to use contraception during the study period and for 6 months after the study period.
* Patients voluntarily joined the study and signed the informed consent, showing good compliance.

Exclusion Criteria:

-Complicated disease and history: A) Has developed other malignant tumors within 2 years or is currently suffering from the same tumor; B) unmitigated toxic reactions above CTC AE grade 1 due to any prior treatment, excluding hair loss and peripheral sensory nerve disorders; C) received major surgical treatment or significant traumatic injury (excluding needle biopsy) within 28 days prior to the commencement of study treatment; D) Long-term unhealed wounds or fractures; E) The occurrence of arterial/venous thrombosis events within 6 months, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism; F) People with a history of psychotropic substance abuse and inability to quit or with mental disorders; G) subjects with any severe and/or uncontrolled disease;"

-Tumor-related symptoms and treatment: A) had undergone surgery, chemotherapy, radiation or other anticancer therapy within 4 weeks prior to the start of study treatment (washout period was calculated from the end of the last treatment); B) Chinese patent drugs with anti-tumor indications specified in the NMPA approved drug specifications (including compound cantharide capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Brucea oil injection/capsule, Xiaoaoping tablet/injection, Huabenin capsule, etc.) were received within 2 weeks before the start of the study; C) previously received immunodouble antibody therapy targeting the same target of TQB2858 injection; D) uncontrolled pleural effusion, pericardial effusion, or ascites that still require repeated drainage (as determined by the investigator); E) Patients with brain metastases whose symptoms stabilized less than 4 weeks after discontinuation of dehydrants and steroids;"

-Research Treatment Related: A) a history of live attenuated vaccine vaccination within 28 days prior to the study treatment initiation or a planned live attenuated vaccine vaccination during the study period; B) Previous history of severe allergy to macromolecular drugs or known components of TQB2858 injection; C) Study the occurrence of active autoimmune disease requiring systemic treatment (e.g., use of palliative drugs, corticosteroids, or immunosuppressants) within 2 years prior to treatment initiation.Alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic; D) have been diagnosed with immunodeficiency or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy.(dose of >10mg/ day prednisone or other equivalent efficacy hormone), and continued to use within 2 weeks of the first administration;" Participants had participated in other antitumor drug clinical trials in the previous 4 weeks;

-Subject who, in the Investigator's judgment, has a concomitant disease that seriously endangers the subject's safety or affects the completion of the study, or is considered unsuitable for inclusion for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Each subject started from the signing of the informed consent until 30 days after the last administration or the start of a new target indication
  The incidence of all adverse events (AE), serious adverse events (SAE) and treatment-related adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Jinlin Cancer Hospital, Changchun, Jilin, China